CLINICAL TRIAL: NCT03764787
Title: A Phase I/II Study of Combination of Hypofractionated Proton Therapy With Immunotherapy
Brief Title: Combination of Hypofractionated Proton Therapy With Immunotherapy
Acronym: I-HypoPT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: YiZhou International Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Xian-shu Gao, Professor, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20181203
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Proton Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation+PD-1 Ab (Experimental): proton radiotherapy concurrent with immunotherapy(ie. PD-1 Ab for 1 year)
  Interventions: Combination Product: Radiation+PD-1 Ab

INTERVENTIONS:
Combination Product: Radiation+PD-1 Ab — combination of proton radiotherapy with PD-1 antibody

SUMMARY:
The purpose of this research study is to compare the effects (good and bad) on subjects and their cancer using hypofractionated proton radiation therapy in combination with immunotherapy(ie. Programmed cell death protein 1, also known as PD-1 antibody). Hypofractionation is a technique that delivers higher daily doses of radiation over a shorter period of time.

DETAILED DESCRIPTION:
Hypofractionated radiotherapy (HFRT), also known as Stereotactic body radiation therapy (SBRT) or Stereotactic ablative radiotherapy (SABR), is a regular pattern of photon radiotherapy. HFRT could achieve comparable curative effect to surgery in variable type of tumor. With the development of proton radiotherapy technology, proton HFRT technique is available nowadays. However, proton HFRT technique is mainly effective in improving the local control rates. This study intends to observe the safety and efficacy of proton HFRT technique combined with immunotherapy in improving the overall anti-tumor effect.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Unspecified Adult Solid Tumor
* Intending to be treated with proton beam and immunotherapy
* Age ≥ 18 years old
* KPS≥70
* Signed written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under guardianship or tutorship
* Patients or legal guardians who are unable to understand informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through 1 years after completion of treatment
  Assess adverse events according to CTCAE4.0

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through 2 years after completion of treatment
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | Through 2 years after completion of treatment
  OS is defined as the duration of time from start of treatment to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Xianshu Gao, MD,PhD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No